CLINICAL TRIAL: NCT03798119
Title: Efficacy and Safety of Switching to Tenofovir Alafenamide for Chronic Hepatitis B Patients With Advanced Fibrosis and Partial Virologic Responses to Oral Nucleos(t)Ide Analogues
Brief Title: TAF Switch in F3/4 CHB pt With Partial Response to NUC (ESTAB-AFPVR)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20180111
Record Dates: First submitted 2018-12-24; First posted 2019-01-09 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2018-12

CONDITIONS: Hepatitis B; Fibrosis and Cirrhosis of Liver
Keywords: Hepatitis B; advanced fibrosis; Cirrhosis; Switch; Tenofovir alafenamide
MeSH Terms: conditions — Hepatitis B; Fibrosis | interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Switch to TAF (Experimental): Subjects who meet the inclusion and exclusion criteria will switch prior NUCs to TAF 25 mg/day for 96 weeks
  Interventions: Drug: Tenofovir Alafenamide

INTERVENTIONS:
Drug: Tenofovir Alafenamide — Subjects in this group will switch prior nucleot(s)ide analogs to Tenofovir Alafenamide 25 mg/day for 96 weeks

SUMMARY:
A total of 80 adult chronic hepatitis B patients with advanced liver fibrosis (including fibrosis stage 3 and cirrhosis), who are currently on nucleot(s)ide analogs (except tenofovir alafenamide) therapy with detectable HBV DNA after 52 weeks of therapy will switch prior NUCs to TAF 25 mg/day for 96 weeks

DETAILED DESCRIPTION:
Study Overview

Dosage regimen: Patients of CHB with advanced fibrosis and partial virological response to NUCs will be considered eligible for the present study. The enrollment will be up to the physician's discretion. The drug will be administered 1 pill (25 mg) per day orally, per manufacturers' instructions, and can be taken with food.

Compliance: Enrolled patients must be monitored according to the protocol, GCP, and clinical practice guidelines.

Study population: Approximately 80 adult CHB patients with advanced fibrosis (including fibrosis stage 3 and cirrhosis), who are currently on NUCs (except TAF) therapy with detectable HBV DNA after 52 weeks of therapy will switch prior NUCs to TAF 25 mg/day for 96 weeks. For patients of fibrosis stage 3, the numbers of enrolled patients will be no more than 40% of total enrolled patients.

Study Objectives

Primary objective:

• To describe the improvement of rate of viral suppression with TAF in patients of partial virological response with previous anti-HBV NUCs.

Secondary objective

* To describe the persistence or improvement of rate of ALT normalization (local and AASLD criteria) with TAF in patients of partial virological response with previous anti-HBV NUCs.
* To describe the trends in serum creatinine, calculated creatinine clearance, and renal tubular function with TAF.
* To describe the trends in bone mineral density with TAF.
* To describe the progression/regression of liver fibrosis with TAF.
* To describe the prespecified factors associated with viral suppression and/or ALT normalization after switching to TAF, including viral resistance profiles, HBsAg levels and HBV viral loads at the initiation of prior NUC and at the time of TAF switching, HBV genotype, hepatic fibrosis, age, sex, prior preparations of NUCs, and host immunogenetics.

Study Procedures:

Pre-Screening: Patients who are currently under HBV NUC, except TAF therapy, with liver fibrosis stage 3 or 4 at the initiation of NUC, and with detectable HBV DNA after week 52 of therapy will be considered eligible in this prospective interventional cohort study. If the patient is deemed eligible to participate, the site will evaluate the potential patient using the inclusion/exclusion criteria and fill out the CRF for the screening visit. The local coordinator will transmit the pre-screening data to the central coordinator prior to the actual screening/baseline visit. If the patient is deemed eligible by the Primary Investigator, the patient will be given a study ID and allowed to enter the study.

Screening/Baseline: Written and informed consent will be obtained prior to any study protocol-related procedures or data abstraction. If the patient has been pre-screened approved and all lab data are available, the participant will begin the study TAF treatment on the screening/baseline visit. The screening/baseline visit consists of obtaining written and informed consent, reviewing the inclusion/exclusion criteria, confirming medical history, completing a physical examination with vital signs and body weight, reviewing any concomitant medications and study drug dispensing. HCV, HDV, and HIV antibody test will be performed after written informed consent is obtained. The samples of HDV antibody test will be collected at local site and sent to KMUH, tested by central lab. Baseline resistance testing will also be performed by direct sequencing.

Procedures: laboratory tests including CBC (complete blood count) panel, Serum Bilirubin (total/direct), AST, ALT, GGT, Albumin, BUN, Creatinine, Na, K, Phosphate, Prothrombin time (INR), and Urine routine/creatinine/phosphate will be done every visit. Pregnant test (only for women of child-bearing potential), Child-Pugh score, and FIB-4 score should also be done every visit. AFP (alpha-fetoprotein), and Abdominal ultrasound should also be done every 3 to 6 months for HCC surveillance. HBV serological markers including HBeAg/HBeAb, HBV DNA quantification (by central lab.) will be done every visit and HBsAg quantification (by central lab.) every 6 months. Bone Density Scan (DEXA) will be done at week 24, 48, and 96. Fibroscan/CAP will be performed at week 48, and 96 to determine regression of fibrosis. Blood will be drawn at the site at which the participant was recruited, and processed by a lab technician in the clinical laboratory at that respective site, except HDV antibody test and HBsAg/HBV DNA quantification which will be performed by the central lab. at KMUH.

Treatment Visits: Treatment will consist of TAF 25 mg daily with food for 96 weeks. Treatment visits will occur at week 4, 12, 24, 36, 48, 72, and 96 as per routine clinical care, except for those who developed virological breakthrough, SAE, or others judged by the investigators. At every visit, the patient must bring all study drugs (including empty bottles), so that the study coordinator can count compliance using the number of remaining pills.

This schedule of clinic visits and laboratory tests are routine and standard practice for investigators in their treatment of similar patients with CHB. Patients will be encouraged to adhere to these recommendations. Results of these laboratory tests and clinical evaluations will be recorded as well as any additional evaluations that are done as part of the patient's clinical care that is pertinent to the objective of the study.

Discontinuation criteria: The study can be terminated at any time for any reasons by Primary Investigator. Though there is no formal treatment stopping rules in this study, patients might be asked to stop if there are any adverse events that the investigator feels make it the patient's best interest to stop treatment.

Withdrawal of Subjects

Withdrawal Criteria:

* Failure to follow study instructions or protocol violation that in the judgment of the investigator
* Serious Adverse Events that in the judgment of the investigator
* Development of virological breakthrough (defined as reappearance of HBV DNA or at least one log10 elevation of HBV DNA from nadir in 2 consecutive measurements one month apart. further treatment plans are at the discretion of the treating physician and patient.
* Any medical, psychosocial or administrative or other reasons that in the judgment of the investigator, be detrimental to the patient's well-being.
* Death
* Withdrawal of informed consent

Adverse Events and Toxicity Management

Assessment of safety: Safety assessments will include monitoring of laboratory results, vital signs, treatment-emergent adverse events, serious adverse events, etc. Safety assessments will be performed at every clinic visit as part of clinical care and during follow-up visits.

If, in Primary Investigator's judgment, a clinical significant worsening from baseline is observed in any laboratory or other test parameters, physical exam finding, or vital sign, a corresponding clinical adverse event should be recorded.

If a specific medical diagnosis has been made, that diagnosis or syndrome should be recorded as the adverse event, whenever possible. However, a complete description of the signs, symptoms, and investigations which led to the diagnosis should be provided. For example, if clinically significant elevations of liver function tests are known to be secondary to hepatitis, "hepatitis" and not "elevated liver function tests" should be recorded. If the cause is not known, the abnormal test or finding should be recorded as an adverse event, using appropriate medical terminology (e/g/ thrombocytopenia, peripheral edema).

Maintenance of Safety Information: Safety information will be maintained in a clinical database/repository in a retrievable format. At a minimum, at the end of the treatment phase (="last patient off treatment") as well as the end of the follow-up phase (="last patient out") of the study, Primary Investigator shall provide all adverse events, both serious and non-serious, in report format.

Statistics

Data management and analysis will be performed at Kaohsiung Medical University Hospital.

Sample size to be used in the analysis: We calculated that a sample size of 80 patients with a 10% dropout rate would provide 85% power to show increased to 30% of virologic response (HBV DNA <LLOQ) rate after 52 weeks of TAF therapy, compared to 15% of continuing prior NUC therapy with a type I error rate of 0.05 for the one-tailed analyses of the primary endpoint.

Statistical methods to be employed: Descriptive and comparative statistics will be performed for all demographic and clinical variables that are outcome endpoints for this pilot study.

Level of significance: A 95% confidence interval will be used.

Termination of trial: Termination of the trial will be upon completion of follow-up of all 80 subjects enrolled and/or up to the discretion of the primary investigator.

Procedure for missing, unused, spurious data: Data that is missing, unused or spurious data will all be treated as missing data. This data will be marked as an empty field.

Deviation from the original statistical plan: Any deviation from the original statistical plan will be up to the discretion of the primary investigator.

Selection of subjects to be included in analyses: All eligible subjects that have not been withdrawn from the study will be included in analyses.

Interim analysis An interim analysis will be performed at Week 24 after all the 80 patients enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥20 years
2. CHB diagnosis confirmed by positive HBsAg or HBV DNA for more than 6 months, or documented history of CHB in medical record before initiation of NUC therapy.
3. Currently maintained on nucleot(s)ide analogues (except TAF) therapy for more than one year, with detectable HBV DNA after 52 weeks of therapy, detectable HBV DNA within 3-6 months prior to screening, and remains detectable HBV DNA at screening.
4. Patients with liver fibrosis stage 3 (defined as Metavir fibrosis stage 3 by liver biopsy, or fibrosis-4 score 3.25 ~ 6.49, or ARFI 1.80 ~ 1.99 m/s, or Fibroscan 9.5~12.4 kPa), or cirrhosis (defined as Metavir fibrosis stage 4 by liver biopsy, or APRI >2, or fibrosis-4 score ≥ 6.5, or ARFI ≥ 2.0 m/s, or Fibroscan ≥12.5 kPa, or image diagnosis with splenomegaly or esophageal/gastric varices) at the initiation of prior NUC therapy or during the prior NUC therapy. The liver biopsy should be within 5 years, or during the prior NUC therapy and other non-invasive assessments should be within 6 months at the initiation of NUC therapy or during the prior NUC therapy.
5. Estimated creatinine clearance > 15 ml/min (using the Cockcroft-Gault method) within 6 months prior to screening. (Note: multiply estimated rate by 0.85 for women).
6. Willing and able to provide informed consent
7. Able to comply with dosing instructions for study drug administration and able to complete the study schedule of assessments

Exclusion Criteria:

1. Pregnant women, women who are breast feeding or who believe they may wish to become pregnant during the course of the study
2. Previous recipient of a liver transplant
3. Co-infection with human immunodeficiency virus (HIV) or hepatitis C (HCV) or hepatitis D (HDV)
4. Severe or uncontrolled comorbidities, determined by the Investigator.
5. Known history of serum albumin level <3 g/dL, or total bilirubin level >3 mg/dL, or presence of ascites.
6. Known history of hepatic encephalopathy, and/or variceal bleeding.
7. Malignancy history including hepatocellular carcinoma, except cancers curable by surgical resection (e.g. basal cell skin cancer and squamous cell cancer within 5 yrs of screening).
8. On any of the disallowed concomitant medications listed in the prior and concomitant medications list (pg. 11). Subjects on prohibited medications who are otherwise eligible will need a wash out period of at least 30 days prior to the Screening.
9. Males and females of reproductive potential who are unwilling to use "effective" protocol-specified method(s) of contraception during the study.
10. Current substance or alcohol abuse judged by the investigator to potentially interfere with subject compliance.
11. Any other clinical conditions that, in the opinion of the Investigator, would make the subject unsuitable or unable to comply with any of the study procedures

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Rate of virological response | at 48 weeks of TAF therapy.
  HBV DNA <LLOQ

SECONDARY OUTCOMES:
Rate of virological response | at 96 weeks of treatment
  HBV DNA <LLOQ
Rate of ALT normalization | at week 48 and 96
  by local (<40 U/L), and AASLD (male ≤35, female ≤25 U/L) criteria
Changes of serum creatinine | at week 48 and 96
Changes of calculated creatinine clearance (Cockcroft-Gault) | at week 48 and 96
Changes in bone mineral density | at week 48 and 96
Changes in liver fibrosis | at week 48 and 96
  determined by Fibroscan

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Lung Yu, Prof., Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No